CLINICAL TRIAL: NCT06931067
Title: Health Behavior Change for Fall Prevention
Brief Title: OTAGO Exercise Program and Motivational Interviewing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Wellness Network (Unknown)
Responsible Party: Principal Investigator, Hiroko Kiyoshi-Teo, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 27787
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Fall Risk Factors; Physical Activity; Engagement, Patient; Community-dwelling Older Adults
Keywords: OTAGO; OEP; Motivational interviewing; behavior change
MeSH Terms: conditions — Motor Activity; Patient Participation | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): OTAGO exercise home visits will be offered 7 times with 2 phone-based check-ins during the 6-month period. As part of OTAGO home visits, participants will receive OTAGO exercise instruction and MI. Each home visit will be approximately an hour.
  Interventions: Behavioral: OTAGO Exercise Program with motivational interviewing

INTERVENTIONS:
Behavioral: OTAGO Exercise Program with motivational interviewing — OTAGO exercise home visits will be offered 7 times with 2 phone-based check-ins during the 6-month period. As part of OTAGO home visits, participants will receive OTAGO exercise instruction and MI. Each home visit will be approximately an hour.

SUMMARY:
The goal of this study is to see if OTAGO instructors, who have been trained in a special communication method called motivational interviewing, can help older adults start and stick with the OTAGO exercise program. The results will help guide future research on how behavior change techniques can support other fall prevention strategies.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the feasibility and impact of OTAGO instructors who are trained in motivational interviewing communication approach to facilitate older adult's uptake of the OTAGO exercises. This study will create the basis for future trials that will explore the impact of behavior change interventions on other fall prevention strategies.

We propose a single-arm quasi-experimental trial with older adults with high fall risks. The study intervention consists of OTAGO visits by study staff (MI-trained OTAGO instructor) over 6 months to improve older adults' engagement in fall prevention behaviors with a focus on OTAGO exercises. Participants will be followed for additional 6 months for the total study duration of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60
* At high fall risk: At least one "Yes" to 1) had a fall in the past year; 2) answer "difficult" to the question "do you find it hard to stand without using your hands"; 3) worry about falling
* Able to converse audibly and coherently in English
* Ambulatory with or without assistive device use
* Self-report challenges navigating the environment outside of the home
* At least one "some or much difficulty" or "unable to do" to:Walking one block?; Stepping up onto a curb?; Getting out of a straight back chair? Climbing one flight of stairs? Getting out of the house

Exclusion Criteria:

* o Receiving ongoing physical therapy with a primary focus on improving balance and strength of lower extremities

  * Experiencing acute health issues such as fracture, pain, or infection that prohibits them from participating in exercises
  * Able to stand on one foot for more than 10 seconds without holding onto something
  * 6-item Callahan cognitive assessment over the phone: Patients with scores of 2 or less, positive for dementia criteria, will be excluded.
  * Patients participating in other studies that may impact fall-related behavior change.
  * Participants engaged in routine moderate or vigorous physical activities that require lower extremity balance and strength (e.g., >100 minutes/week for more than 3 months)

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
OTAGO exercise adherence | Baseline, 6-months & 12 months
  Number of instructed OTAGO exercises completed in a week

SECONDARY OUTCOMES:
4-stage balance test | Baseline & 6-months
  Participants are asked to hold four standing positions that get progressively harder to maintain.
  1. Stand with your feet side-by-side
  2. Place the instep of one foot so it is touching the big toe of the other foot.
  3. Tandem stance Place one foot in front of the other, heel touching toes
  4. Stand on one foot.
Sit-to-stand test | Baseline & 6-months
  Participants are asked to stand from a seated position. We count the number of sit-stand-sit repetitions completed during 30 seconds
Falls Efficacy Scale Short International | Baseline, 6-months, and 12-months
  Measures levels of concern about falls. 7-item, 4-point Likert-type scale; 28: highest concern

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study IPD may be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the completion of all study data collection, analysis, and publication. IPD will be available for 5 years.
Access Criteria: Individuals interested in IPD must contact the PI.